CLINICAL TRIAL: NCT06175208
Title: Targeting Fear of Cancer Recurrence in Cancer Survivors: a Multicentre Randomized Controlled Trial to Evaluate Internet-Based Emotional Freedom Techniques and Internet-Based Mindfulness Meditation as Intervention Strategies
Brief Title: Targeting Fear of Cancer Recurrence in Cancer Survivors: Evaluation of Internet-Based Emotional Freedom Techniques and Internet-Based Mindfulness Meditation as Intervention Strategies
Acronym: REMOTE
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: General Hospital Groeninge (Other)
Collaborators: Kom Op Tegen Kanker (Other); az Glorieux (Unknown); AZ Klina (Other); AZ Vesalius (Other); Imeldaziekenhuis (Other); Jessa Hospital (Other); University Hospital, Antwerp (Other); Universitair Ziekenhuis Brussel (Other); University Hospital, Ghent (Other); Universitaire Ziekenhuizen KU Leuven (Other); Vitaz (Other)
Responsible Party: Principal Investigator, Dr. Philip Debruyne, Principal Investigator, General Hospital Groeninge
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 23435_ REMOTE
Record Dates: First submitted 2023-11-21; First posted 2023-12-18 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Fear of Cancer Recurrence
Keywords: Fear of Cancer Recurrence; Emotional Freedom Techniques; Mindfulness Meditation; Cancer survivors; Psychosocial cancer-related symptoms
MeSH Terms: interventions — Mindfulness

STUDY DESIGN:
Intervention Model Description: This is a multi-site, randomized, three arm trial that will evaluate the efficacy of two distinct types of group interventions to target fear of cancer recurrence (FCR) in cancer survivors.
  The first intervention entails emotional freedom techniques (EFT). The other intervention is mindfulness meditation. The third group is the wait-list control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- internet-based Emotional Freedom Techniques (iEFT) (Experimental): The first intervention entails emotional freedom techniques (EFT). EFT is a brief and easy to learn exposure therapy, originally developed to manage phobias and nowadays known to have many positive effects on both physiological and psychological aspects. Participants will apply EFT daily for the period of 6 weeks. During the trajectory, there is a first information session for participants (±20 minutes) and two follow-up sessions (±15 minutes). These sessions will be guided by the iEFT practitioner. This is an oncology health professional who has gone through a specific EFT training acknowledged by EFT International and is thus qualified and trained to conduct the trial.
  Interventions: Behavioral: Emotional Freedom Techniques
- internet-based mindfulness meditation intervention (iMMI) (Active Comparator): The second intervention is a mindfulness meditation-based intervention focused on improving psychological, behavioural, and biological function in cancer survivors based on following sources: Mindfulness trainingsboek, Het achtweekse programma, stap voor stap (1), Mindfulness bij stress, burn-out en depressie, Een 8-weken-stappenplan voor hulpverleners (2), Mindfulness-based cognitive therapy for depression (3), Met radicale compassie naar de wereld kijken, De RAIN-methode (4). The mindfulness group intervention programme will be conducted once a week, for 2 hours during 6 weeks, by a trained mindfulness provider who will follow the study intervention protocol. Participants will apply mindfulness meditation daily for the period of 6 weeks.
  Interventions: Behavioral: Mindfulness Meditation
- Wait-list Control Group (WLC) (No Intervention): The third arm of the study refers to the wait-list control (WLC) group with delayed intervention offered to the participants after they have completed parallel outcome assessments alongside the participants receiving the two interventions iEFT and iMMI, but not until the end of data collection (i.e. 6 weeks after the post-intervention assessment T1 for the cohort). Patients included in the WLC group can optionally join either the iEFT or iMMI group according to their preference, after 12 weeks (T2).

INTERVENTIONS:
Behavioral: Emotional Freedom Techniques — Every participant may be randomized to either the iEFT, iMMI, or WLC group. All patients will be randomised to one of the three groups and be involved in a 6-week trajectory.
  Other Names: iEFT
  Arms: internet-based Emotional Freedom Techniques (iEFT)
Behavioral: Mindfulness Meditation — Every participant may be randomized to either the iEFT, iMMI, or WLC group. All patients will be randomised to one of the three groups and be involved in a 6-week trajectory.
  Other Names: iMMI
  Arms: internet-based mindfulness meditation intervention (iMMI)

SUMMARY:
In this trial, the investigators introduce two internet-based psychological methods to meet the currently unmet medical need to cope with Fear of Cancer Recurrence (FCR) beyond the acute phase of cancer treatment: internet-based emotional freedom techniques (iEFT) and internet-based mindfulness intervention (iMMI). The primary aim of this trial is to examine the efficacy of Internet-Based Emotional Freedom Techniques (iEFT) and Internet-Based Mindfulness Meditation Intervention (iMMI) to alleviate Fear of Cancer Recurrence (FCR) in cancer survivors, as determined through the Fear of Cancer Recurrence Inventory (FCRI) in cancer survivors. To translate a statistically significant effect on FCR into a clinically significant change, the investigators would need to detect a between-group difference in mean FCRI at T1 of 10 points using an independent samples t-test (two experimental groups are compared against a single wait-list control). When the application of iEFT and/or iMMI appears effective to reduce FCR, these self-help methods could be implemented in clinical settings. The use of these low cost interventions with a low threshold, by an internet-based approach, will facilitate a potential implementation in clinical practice.

DETAILED DESCRIPTION:
Despite our adequate medical care and financial support systems, the mental wellbeing and quality of life after cancer diagnosis and treatment is often poorly addressed in clinical settings. Previous research showed that Fear of Cancer Recurrence (FCR) is one of the most common psychological burdens faced by 39%-97% of cancer survivors. In this phase III randomized multicentre trial, patients will be allocated to either the iEFT group, iMMI group or wait-list control (WLC) group for a study trajectory of 6 weeks. 339 cancer survivors, between 6 months and 5 years since diagnosis, and who have completed their primary cancer treatment (i.e. surgery, radiation, and/or chemotherapy) will be enrolled and randomized 1:1:1 to one of the two intervention groups or the WLC group. Participants will complete evaluation questionnaires at baseline (T0), after 6 weeks (T1) and 12 weeks (T2) of intervention or waiting list, and 24 weeks (T3). A biomarker endpoint includes the measurement of chronic biologic stress in hair cortisol concentration. Therefore, optional hair collection may take place before (T0) and after the 6-week intervention (T1). Primary objective is to evaluate the feasibility and efficacy of iEFT and iMMI as an intervention strategy to reduce FCR in cancer survivors. The investigators hypothesize that an intervention with iEFT or iMMI will be superior compared to the WLC group at T1. Secondary objectives include the following:

ELIGIBILITY:
Inclusion Criteria:

* Patients should have reached a minimum age of 18 years at the time of enrolment
* Patients should have a histologically confirmed diagnosis of a solid cancer or haematologic malignancy
* Patients should have completed surgery, chemotherapy, radiation therapy, immunotherapy, hormone therapy, targeted drug therapy or a combination of these at least 2 months ago and no longer than 5 years ago at the time of enrolment
* Patients should have an expected life expectancy of at least 5 years
* Patients are disease-free at the time of enrolment, as defined by the absence of somatic disease activity parameters
* Patients can be included in a stable phase of their immunotherapy (e.g. adjuvant use of checkpoint inhibitors for melanoma), hormonal therapy (e.g. for breast and prostate cancer), targeted drug therapy (e.g. trastuzumab and pertuzumab for breast cancer; stable dose of PARP inhibitors for ovarian cancer; retuximab for lymphoma), or a combination of these
* Patients must suffer from high FCR based on the Cancer Worry Scale (cut-off ≥ 14)
* Patients should be able to adequately communicate in Dutch
* Patients should present with a sufficient mental and physical functional status (according to investigator's judgment and first baseline assessment) for completing the questionnaires and neuropsychological assessment
* Patients under current treatment for a depression or anxiety disorder are allowed to enrol provided their depression or anxiety disorder is stable

Exclusion Criteria:

* Patients who received a treatment with palliative intent
* Patients showing signs of mental deterioration
* Patients suffering from organic brain syndrome (concussion without neurological symptoms and negative imaging is allowed)
* Patients who are alcohol or drug dependent
* Patients with another serious or chronic medical, neurologic or psychiatric condition that contributes to substantial physical or emotional disability that would detract from participating in either of the intervention programmes or from the measurement of intervention outcomes; a prior diagnosis of a depressive, anxiety or adjustment disorder is allowed
* Patients who cannot commit to the intervention schedule; obstacles such as surgery or long-term hospitalisation, change of residence or work, … can have an emotional and practical impact which makes these patients not eligible for participation.
* Patients who actively practice EFT or mindfulness(based) meditation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 339 (Estimated)
Dates: Start 2024-07-03 (Actual); Primary Completion 2028-08-01 (Estimated); Study Completion 2028-10-30 (Estimated)

PRIMARY OUTCOMES:
Fear of Cancer Recurrence | 6 weeks (T1)
  The primary endpoint will be reached after the first period of performing iEFT or iMMI during 6 weeks or be at the waiting list for 6 weeks (T1) where we will look at the efficacy of iEFT and iMMI to alleviate of Fear of Cancer Recurrence (FCR) based on the Fear of Cancer Recurrence Inventory (FCRI). FCRI has a minimum value of 0 and maximum value of 168, with a higher score pointing out to a worse outcome.

SECONDARY OUTCOMES:
Follow-up of Fear of Cancer Recurrence | T0 (baseline), T1 (6 weeks), T2 (12 weeks) and T3 (24 weeks)
  Efficacy of iEFT and iMMI to reduce FCR (Fear of Cancer Recurrence Inventory; FCRI). FCRI has a minimum value of 0 and maximum value of 168, with a higher score pointing out to a worse outcome.
Psychological Distresss | T0 (baseline), T1 (6 weeks), T2 (12 weeks) and T3 (24 weeks)
  Efficacy of iEFT and iMMI to reduce psychological distress (Distress Thermometer). Distress thermometer has a minimum value of 0 and maximum value of 10, with a higher score pointing out to a worse outcome.
Psychological Distresss | T0 (baseline), T1 (6 weeks), T2 (12 weeks) and T3 (24 weeks)
  Efficacy of iEFT and iMMI to reduce psychological distress (38-item Problem list). The Distress Thermometer includes 36 problems answered with "no" or "yes" clustered into five domains: practical problems, family problems, emotional problems, spiritual problems, and physical problems.
Fear of Cancer Recurrence | T0 (baseline), T1 (6 weeks), T2 (12 weeks) and T3 (24 weeks)
  Efficacy of iEFT and iMMI to enhance Quality of Life (EORTC QOL Cancer Survivorship Core Questionnaire (QLQ-SURV100), amended with items from the EORTC Core QOL questionnaire QLQ-C30). EORTC QLQ-SURV 100 has a minimum value of 100 and maximum value of 406, with a higher score pointing out to a better outcome. EORTC QLQ-C30 has a minimum value of 30 and maximum value of 126, with a higher score pointing out to a better outcome.
Fear of Cancer Recurrence | T0 (baseline), T1 (6 weeks), T2 (12 weeks) and T3 (24 weeks)
  Efficacy of iEFT and iMMI to enhance health status (EuroQol EQ-5D-5L). The visual analogue scale of the EuroQol EQ-5D-5L has a minimum value of 0 and maximum value of 100, with a higher score pointing out to a better outcome.
Number of participants continuing the intervention after T1 | T2 (12 weeks) and T3 (24 weeks)
  To identify the continuous application of iEFT or iMMI, participants will need to answer the questionnaire about whether they cotinue the application of EFT or mindfulness meditation, and the frequency of application, post-intervention period.

OTHER OUTCOMES:
Biomarker endpoint | T0 (baseline), T1 (6 weeks), but this endpoint will be completed only when the primary objective would be positive at T1
  • Effect of iEFT and iMMI on chronic biological stress measure as hair cortisol concentration

CONTACTS AND LOCATIONS:
Overall Officials: Philip R Debruyne, MD, PhD, Principal Investigator — Kortrijk Cancer Centre,General Hospital Groeninge
Locations (11):
- Belgium (11):
  - AZ Klina, Brasschaat, Antwerp
  - University Hospital Antwerp, Edegem, Antwerp
  - University Hospital Gent, Ghent, East-Flanders
  - University Hospital Leuven, Leuven, Vlaams-Brabant
  - Kortrijk Cancer Centre, az groeninge, Kortrijk, West-Flanders
  - Imelda ziekenhuis, Bonheiden
  - Jessa ziekenhuis, Hasselt
  - University Hospital Brussels, Jette
  - AZ Glorieux, Ronse
  - VITAZ, Sint-Niklaas
  - AZ Vesalius, Tongeren

IPD SHARING:
Plan to Share IPD: No
At the moment, there is no plan to make individual participant data (IPD) available to other researchers. Moreover, data will be pseudonimyzed.

REFERENCES:
- [Result] Tack L, Lefebvre T, Lycke M, Langenaeken C, Fontaine C, Borms M, Hanssens M, Knops C, Meryck K, Boterberg T, Pottel H, Schofield P, Debruyne PR. A randomised wait-list controlled trial to evaluate Emotional Freedom Techniques for self-reported cancer-related cognitive impairment in cancer survivors (EMOTICON). EClinicalMedicine. 2021 Aug 19;39:101081. doi: 10.1016/j.eclinm.2021.101081. eCollection 2021 Sep. PMID 34466793